CLINICAL TRIAL: NCT04280874
Title: Comparison of Intracervical and Intravaginal Application of Prostaglandin E2 for Induction of Labour in Term Pregnancies With Unfavourable Cervix
Brief Title: Induction of Labor in Term Pregnancies With Unfavourable Cervix
Acronym: RAND
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Merkur (Other)
Responsible Party: Principal Investigator, Katja Vince, Principal Investigator, Clinical Hospital Merkur
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RANDOM1
Record Dates: First submitted 2020-02-14; First posted 2020-02-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Induction of Labor Affected Fetus / Newborn; Prostaglandins Causing Adverse Effects in Therapeutic Use
Keywords: dinoprostone; Bishop score; labor induction; term pregnancy
MeSH Terms: interventions — Dinoprostone; KLK15 protein, human

STUDY DESIGN:
Intervention Model Description: 212 pregnant women are randomly assigned into 2 groups for application of one of two dinoprostone agents used for labor induction (intravaginal or intracervical dinoprostone)
Who Masked: Participant
Masking Description: two dinoprostone agents are randomly applied and compared - one in patient's cervix and the other in vagina without the patient knowing which agent is applied
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Active Comparator): 106 randomly selected pregnant women
  Interventions: Drug: Dinoprostone 0.5 MG
- GROUP B (Active Comparator): 106 randomly selected pregnant women
  Interventions: Drug: Dinoprostone 2 MG/2.5 ML Vaginal Gel/Jelly

INTERVENTIONS:
Drug: Dinoprostone 0.5 MG — 0.5mg dinoprostone applied intracervically
  Other Names: PREPIDIL
  Arms: GROUP A
Drug: Dinoprostone 2 MG/2.5 ML Vaginal Gel/Jelly — 2mg dinoprostone applied intravaginally
  Other Names: PROSTIN
  Arms: GROUP B

SUMMARY:
This is a prospective randomized trial comparing two prostaglandin E2 (dinoprostone) agents used for labor induction in pregnant women with term pregnancies and unfavorable cervix.

DETAILED DESCRIPTION:
This prospective randomized trial includes pregnant women with term pregnancies, indication for labor induction and an unfavorable cervix. These women are randomized into two groups: one group is induced using an intracervical prostaglandin E2 (PGE2, dinoprostone) formulation, the other using an intravaginal PGE2 formulation. Main outcome is time period between beginning of labor induction to delivery, and a reduction of four hours is considered clinically significant.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancies (> 37 weeks gestation)
* unfavourable cervix (Bishop score <6)
* indication for labor induction
* absence of uterine contractions
* reassuring cardiotocography

Exclusion Criteria:

* ruptured membranes
* scar uterus (previous caesarean section or uterus surgery)
* pregnancy complications: intrauterine growth restriction; oligohydramnios, pre-eclampsia, non-reassuring/pathological cardiotocography, cholestasis in pregnancy, diabetes mellitus, multifetal pregnancy, breech presentation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
time period between beginning of labor induction to delivery | 5 days
  hours (difference of 4 hours or more is considered significant)

SECONDARY OUTCOMES:
number of births within 24h of start of labor induction | 7 days
  N (%)
number of deliveries by caesarean section or instrumental deliveries | 7 days
  N (%)
number of uterus hyperstimulation | 7 days
  N (%)

CONTACTS AND LOCATIONS:
Overall Officials: Katja Vince, MD, Study Chair — Clinical Hospital Merkur
Locations (1):
- Clinical Hospital Merkur, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No